CLINICAL TRIAL: NCT07318129
Title: Indole-3-PROpionic Acid Clinical Trials - Multiple Sclerosis (iPROACT-MS)
Brief Title: Indole-3-PROpionic Acid Clinical Trials - Multiple Sclerosis
Acronym: iPROACT-MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: University of Copenhagen (Other); University of Southampton (Other)
Responsible Party: Principal Investigator, Jette Lautrup Frederiksen, MD, dr.med, professor at DMSc, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-25042489
Record Dates: First submitted 2025-11-23; First posted 2026-01-05 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Relapsing Remitting Multiple Sclerosis (RRMS)
Keywords: indole-3-propionic acid; multiple sclerosis; gut bacterial metabolite; dietary supplement; gut-brain axis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each set of capsule containers (the containers to be used by a study participant during the intervention) is labelled with a unique ID and no other identifier. A randomization key is prepared by an external party randomizing study participants to IPA or placebo using stratified block randomization with random block sizes of 4 or 6. Stratification accounts for recent evidence of disease activity (yes vs. no) defined as experience of clinical relapses within the past year or demonstration of new, contrast-enhanced or enlarged lesions on a clinical MRI scan performed within the last 12 months from randomization.
  A software system is used to reveal the unique container ID to be used by each randomized participant without revealing its corresponding arm. Only after all study participants have completed the trial and the collected data have been cleaned and quality checked, are the researchers performing the statistical analyses informed about which participants belong to each arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsules
  Interventions: Dietary Supplement: Placebo
- Indole-3-propionic acid (IPA) (Experimental): IPA capsules
  Interventions: Dietary Supplement: Indole-3-propionic acid (IPA)

INTERVENTIONS:
Dietary Supplement: Placebo — Two capsules are taken every morning and two capsules are taken every evening for 27 consecutive months. Placebo capsules are taken orally.
  Arms: Placebo
Dietary Supplement: Indole-3-propionic acid (IPA) — Two capsules are taken every morning and two capsules are taken every evening for 27 consecutive months. Active capsules are taken orally and contain 250 mg of IPA each resulting in a total daily dose of 1000 mg of IPA.
  Arms: Indole-3-propionic acid (IPA)

SUMMARY:
This study, iPROACT-MS, is part of the iPROACT group of clinical trials aiming to investigate the effects of oral supplementation with indole-3-propionic acid (IPA) in humans. IPA is naturally produced as a gut bacterial metabolite with the amino acid tryptophan as substrate. The primary aim of iPROACT-MS is to investigate whether patients with relapsing-remitting multiple sclerosis (RRMS) can benefit from supplementation with IPA. The hypothesis is that supplementation with IPA will protect against MS-related disease activity, neurodegeneration and metabolic abnormalities. Secondary, iPROACT-MS aims at elucidating the complex relationships between lifestyle, gut microbial factors, inflammation, oxidative stress, metabolic health, MS disease severity and MS disease activity.

ELIGIBILITY:
Inclusion Criteria:

* Women and men ≥18 and ≤65 years of age
* Diagnosed with RRMS according to the 2017 McDonald criteria (or newer updates)
* Routinely treated and monitored for MS
* Speak and read Danish
* Deemed physically and mentally able to participate in this study

Exclusion Criteria:

* Active malignancy
* Diagnosis of Crohn's disease and ulcerative colitis
* Other comorbidities deemed to be relevant
* Haematopoietic stem cell transplantation
* Current or past treatment with non-MS related treatments deemed to be relevant
* Pregnancy or lactation
* People with MR contraindications:

  * Severe claustrophobia
  * Incompatible implants/ foreign objects, including implanted pacemakers, heart valve prostheses, prostheses in the middle ear, implanted devices (e.g., insulin pump), metal debris, e.g., metal splinters in the eyes, miscellaneous shunts and catheters, metal clips from operations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2028-07-15 (Estimated); Study Completion 2028-07-15 (Estimated)

PRIMARY OUTCOMES:
No evidence of disease activity (NEDA) | The time between month 3 and month 27 after initiation of supplementation.
  The percentage of patients that maintain no evidence of disease activity (NEDA-3) in the time between month 3 and month 27 after initiation of supplementation. NEDA-3 is defined as a binary composite consisting of absence of confirmed relapses, no new or enlarged lesions on brain MRI and no confirmed disability progression. For relapses to be confirmed, they need to be accompanied by an increase of at least 0.5 points on the EDSS or 2 points in one of the EDSS functional system scores, or at least 1 point in two or more of the EDSS functional system scores. Confirmed disability progression is defined as an increase in the EDSS score compared to EDSS at month 3 which is of at least 1 point (or 0.5 points if the baseline EDSS >5.5) and is sustained for three months (measured at month 12 and confirmed at month 15 or measured at month 24 and confirmed at month 27 or measured at a relapse evaluation prior to or at month 24 and confirmed at the next visit or the latest at month 27).

SECONDARY OUTCOMES:
Annualized relapse rate evaluated at month 27 | The time between month 3 and month 27 after initiation of supplementation.
  Defined as the total number of confirmed relapses experienced during the intervention for each patient divided by years of exposure to the intervention and excluding the first three months for both outcome and exposure.
Total (cumulative) number of new or enlarged T2-weighted/FLAIR brain lesions per scheduled yearly MRI evaluated at month 27 | The time between month 3 and month 27 after initiation of supplementation.
  New or enlarged brain lesions are evaluated at month 15 and compared to month 3 and at month 27 and compared to month 15; results from unscheduled MRIs between month 3 and month 27 are also considered.
Serum neurofilament light chain (sNfL) | Evaluated longitudinally at months 0, 3, 15 and 27.
Percentage of patients with disability improvement confirmed at 3 months | The time between month 3 and month 27 after initiation of supplementation.
  Confirmed disability improvement is defined as a reduction in EDSS (expanded disability status scale) score compared to EDSS at month 3 which is of at least 1 point (or 0.5 points if the baseline EDSS >5.5). The EDSS score ranges from 0 to 10 with 0 indicating no neurological disability and 10 indicating death from MS. Measured at month 12 and confirmed at month 15 or measured at month 24 and confirmed at month 27.
The time to onset of disability worsening confirmed at 3 months | The time between month 3 and month 27 after initiation of supplementation.
  Confirmed disability worsening is defined as an increase in the EDSS (expanded disability status scale) score compared to EDSS at month 3 which is of at least 1 point (or 0.5 points if the baseline EDSS >5.5). The EDSS score ranges from 0 to 10 with 0 indicating no neurological disability and 10 indicating death from MS. Measured at month 12 and confirmed at month 15 or measured at month 24 and confirmed at month 27 or measured at a relapse evaluation prior to or at month 24 and confirmed at the next visit or the latest at month 27.
Cumulative change in EDSS score | The time between month 3 and month 24 after initiation of supplementation.
  Calculated as area under the curve (AUC) for measured values of the EDSS (expanded disability status scale) score from month 3 to month 24. The EDSS score ranges from 0 to 10 with 0 indicating no neurological disability and 10 indicating death from MS.
Multiple Sclerosis Functional Composite (MSFC) | The time between month 0 and month 24 after initiation of supplementation.
  A composite score used to assess neurological function by combining results from the Timed 25-Foot Walk (T25FW) test, the Nine-Hole Peg Test (9HPT) and the Symbol Digit Modalities Test (SDMT) evaluated at months 0, 12 and 24.
Symbol Digit Modalities Test (SDMT) | The time between month 0 and month 24 after initiation of supplementation.
  A measure of cognitive function and especially processing speed - evaluated at months 0, 12 and 24.
California Verbal Learning Test-II (CVLT-II) | The time between month 0 and month 24 after initiation of supplementation.
  A measure of verbal learning and memory - evaluated at months 0, 12 and 24.
Brief Visuospatial Memory Test - Revised (BVMR-R) | The time between month 0 and month 24 after initiation of supplementation.
  A measure of visuospatial memory - evaluated at months 0, 12 and 24.
Intra-eye change in peripapillary retinal nerve fiber layer (RNFL) thickness | The time between month 0 and month 24 after initiation of supplementation.
  Measured using Optical Coherence Tomography (OCT) at months 0, 12 and 24.
Intra-eye change in ganglion cell and inner plexiform layer (GCIPL) thickness | The time between month 0 and month 24 after initiation of supplementation.
  Measured using Optical Coherence Tomography (OCT) at months 0, 12 and 24.
Modified Fatigue Impact Scale (MFIS-21) | The time between month 0 and month 24 after initiation of supplementation.
  The MFIS-21 consists of a physical subscale (ranges from 0-36), a cognitive subscale (ranges from 0-40) and a psychosocial subscale (ranges from 0-8). The total MFIS-21 scale is computed by adding the scores from the physical, the cognitive and the psychosocial subscales. It ranges from 0-84 with higher scores indicating a greater impact from fatigue. MFIS-21 is evaluated longitudinally at months 0, 3, 6, 9, 12, 15, 18, 21, 24 and 27.
Multiple Sclerosis Quality of Life-54 (MSQOL-54) | The time between month 0 and month 24 after initiation of supplementation.
  The MSQOL-54 questionnaire is used to calculate a physical health composite score and a mental health composite score. They both range from 0-100 with higher scores indicating better health/ higher quality of life. The questionnaire is administered at months 0, 12 and 24.
Brain-derived neurotrophic factor (BDNF) | The time between month 0 and month 27 after initiation of supplementation.
  Brain-derived neurotrophic factor measured in platelet-free plasma samples using ELISA or mesoscale. Monitored longitudinally at months 0, 3, 15 and 27.
C-reactive protein (CRP) | The time between month 0 and month 27 after initiation of supplementation.
  CRP measured in plasma (mg/L) as a biomarker of infection and systemic inflammation. Lower-limit of quantification: 0,4 mg/L. Values below 0,4 mg/L are imputed as 0,2 mg/L. Monitored longitudinally at months 0, 3, 15 and 27.
Triglycerides | The time between month 0 and month 27 after initiation of supplementation.
  Plasma triglycerides (mmol/l) monitored longitudinally at months 0, 3, 15 and 27.
Non-HDL cholesterol | The time between month 0 and month 27 after initiation of supplementation.
  Non-HDL cholesterol calculated as total cholesterol minus HDL cholesterol (mmol/l). Monitored longitudinally at months 0, 3, 15 and 27.
C-peptide | The time between month 0 and month 27 after initiation of supplementation.
  Proinsulin C-peptide (pmol/l) measured in plasma. Monitored longitudinally at months 0, 3, 15 and 27.
Fasting glucose | The time between month 0 and month 27 after initiation of supplementation.
  Plasma glucose (mmol/l). Participants abstain from eating and drinking after 22.00 the day before. Only water is allowed. Monitored longitudinally at months 0, 3, 15 and 27.
8-iso-prostaglandin F2α and other F2-isoprostanes | The time between month 0 and month 27 after initiation of supplementation.
  F2-isoprostanes with a specific focus on 8-iso-prostaglandin F2α measured in morningurine or blood samples as a marker of oxidative stress-related lipid oxidation. Monitored longitudinally at months 0, 3, 15 and 27.
8-oxo-dG | The time between month 0 and month 27 after initiation of supplementation.
  8-oxo-dG (8-Oxo-2'-deoxyguanosine) measured in blood or morningurine samples as a marker of oxidative stress-related DNA damage. Monitored longitudinally at months 0, 3, 15 and 27.
Fecal lipocalin | The time between month 0 and month 27 after initiation of supplementation.
  Lipocalin measured in fecal samples as a sensitive biomarker of intestinal inflammation. Monitored longitudinally at months 0, 3, 15 and 27.
Microbiota profiling of fecal samples | The time between month 0 and month 27 after initiation of supplementation.
  Microbiota profiling of fecal samples using molecular biology methods including but not limited to sequencing and flowcytometric analyses. Monitored longitudinally at months 0, 3, 15 and 27.
Serum and fecal metabolomics | The time between month 0 and month 27 after initiation of supplementation.
  Targetted and untargetted liquid-chromatography mass-spectrometry-based metabolomics to measure diet-, host- and microbial-derived metabolites. Targetted analyses aim to quantify indole-3-propionic acid and its metabolites (biomarker of compliance as well as absorptive and metabolic capacity), other bacterial- and host metabolites of tryptophan as well as short-chain fatty acids. Monitored longitudinally at months 0, 3, 15 and 27.

OTHER OUTCOMES:
Percentage of patients with progression independent of relapse and/or MRI activity | The time between month 3 and month 24 after initiation of supplementation.
  Tertiary efficacy outcome related to multiple sclerosis. Progression is defined as an increase in the EDSS score compared to the EDSS at month 3 which is of at least 1 point (or 0.5 points if the baseline EDSS >5.5). The EDSS score ranges from 0 to 10 with 0 indicating no neurological disability and 10 indicating death from MS. Measured at month 12 and confirmed at month 15 or measured at month 24 and confirmed at month 27.
Six Spot Step Test (SSST) | The time between month 0 and month 24 after initiation of supplementation.
  Tertiary efficacy outcome related to multiple sclerosis. A measure of walking ability, including speed, co-ordination and balance - evaluated at month 0, month 12 and month 24.
Nine-Hole Peg Test (9-HPT) | The time between month 0 and month 24 after initiation of supplementation.
  Tertiary efficacy outcome related to multiple sclerosis. A measure of finger dexterity - evaluated at months 0, 12 and 24.
Glial Fibrillary Acidic Protein (GFAP) | The time between month 0 and month 27 after initiation of supplementation.
  Tertiary efficacy outcome related to multiple sclerosis. Monitored longitudinally in serum samples at months 0, 3, 15 and 27.
Chitinase 3 Like 1 (CHI3L1) | The time between month 0 and month 27 after initiation of supplementation.
  Tertiary efficacy outcome related to multiple sclerosis. Monitored longitudinally in serum samples at months 0, 3, 15 and 27.
Chitotriosidase 1 (CHIT1) | The time between month 0 and month 27 after initiation of supplementation.
  Tertiary efficacy outcome related to multiple sclerosis. Measured longitudinally in serum samples at months 0, 3, 15 and 27.
Work Productivity and Activity Impairment (WPAI) questionnaire | The time between month 0 and month 24 after initiation of supplementation.
  Tertiary efficacy outcome related to multiple sclerosis. WPAI results are expressed as impairment percentages where higher percentages indicate greater impairment and lower productivity. Evaluated at months 0, 12 and 24.
Glycated hemoglobin (HbA1c) | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome related to metabolic health. HbA1c (IFCC, mmol/mol) measured in whole blood. Estimated average glucose values (mmol/l) are also calculated automatically from HbA1c by our laboratory. Monitored longitudinally at months 0, 3, 15 and 27.
Total cholesterol | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome related to metabolic health. Plasma cholesterol (mmol/l). Monitored longitudinally at months 0, 3, 15 and 27.
HDL cholesterol | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome related to metabolic health. Plasma high-density lipoprotein (HDL) (mmol/l). Monitored longitudinally at months 0, 3, 15 and 27.
LDL cholesterol | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome related to metabolic health. Plasma low-density lipoprotein (LDL) (mmol/l). Monitored longitudinally at months 0, 3, 15 and 27.
VLDL cholesterol | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome related to metabolic health. Plasma very low-density lipoproteins (mmol/l). Monitored longitudinally at months 0, 3, 15 and 27.
Body mass index (BMI) | The time between month 0 and month 24 after initiation of supplementation.
  Exploratory outcome related to metabolic health. BMI calculated as weight (kg)/ height (m)^2. Monitored longitudinally at months 0, 12, and 24. Height is only measured at baseline with longitudinal changes in BMI reflecting changes in weight.
Sagittal abdominal diameter (SAD) | The time between month 0 and month 24 after initiation of supplementation.
  Exploratory outcome related to metabolic health. The distance (cm) from the lower back to the highest point of the abdomen while in a supine position as a measure of visceral obesity. Monitored longitudinally at months 0, 12 and 24.
Waist circumference | The time between month 0 and month 24 after initiation of supplementation.
  Exploratory outcome related to metabolic health. Calculated as an average of two measurements and expressed in cm. Monitored longitudinally at months 0, 12 and 24.
Hip circumference | The time between month 0 and month 24 after initiation of supplementation.
  Exploratory outcome related to metabolic health. Calculated as an average of two measurements and expressed in cm. Monitored longitudinally at months 0, 12 and 24.
Waist-to-Hip ratio | The time between month 0 and month 24 after initiation of supplementation.
  Exploratory outcome related to metabolic health. Monitored longitudinally at months 0, 12 and 24.
Blood pressure | The time between month 0 and month 24 after initiation of supplementation.
  Exploratory outcome related to metabolic health. Blood pressure (mm Hg) defined as the lowest value obtained across three measurements. Monitored longitudinally at months 0, 12 and 24.
Resting heart rate | The time between month 0 and month 24 after initiation of supplementation.
  Exploratory outcome related to metabolic health. Resting heart rate defined as the lowest value obtained across three measurements while sitting in a relaxed position. Monitored longitudinally at month 0, 12 and 24.
Flowcytometric analyses of microvesicles and endothelial progenitor cells | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome related to systemic inflammation. Monitored longitudinally in platelet-free plasma at months 0, 3, 15 and 27.
Circulating cytokines and acute phase reactants | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome related to systemic inflammation. Monitored longitudinally at months 0, 3, 15 and 27.
Serum antibodies | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome related to systemic inflammation. Monitored longitudinally at months 0, 3, 15 and 27.
Urinary neopterin | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome related to systemic inflammation. Monitored longitudinally at months 0, 3, 15 and 27.
suPAR | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome related to systemic inflammation. Soluble urokinase plasminogen activator receptor (suPAR) monitored longitudinally in blood samples at months 0, 3, 15 and 27.
Osteopontin | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome related to systemic inflammation. Monitored longitudinally in blood samples at months 0, 3, 15 and 27.
Buffycoat gene expression analyses | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome related to systemic inflammation. Gene expression analyses monitored longitudinally in buffycoat samples collected at months 0, 3, 15 and 27.
Protein carbonyls | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome related to oxidative stress. Protein carbonyls measured in blood or morningurine samples as a marker of protein oxidation. Monitored longitudinally at months 0, 3, 15 and 27.
Malondialdehyde | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome related to oxidative stress. Malondialdehyde monitored longitudinally in blood or morningurine samples at months 0, 3, 15 and 27.
Glial cell line-derived neurotrophic factor (GDNF) | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome monitored longitudinally at months 0, 3, 15 and 27.
Platelet-derived growth factor (PDGF) | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome monitored longitudinally at months 0, 3, 15 and 27.
Gastrointestinal comfort and bowel movement pattern | The time between month 0 and month 24 after initiation of supplementation.
  Exploratory outcome related to gastrointestinal function. Self-reported (questionnaire) gastrointestinal symptoms of bloating, pain, rumbling, flatulence, constipation, hard stools and diarrhea evaluated using a visual analogue scale as well as a question on the frequency of defecation. Monitored longitudinally at months 0, 12 and 24.
Stool consistency | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome related to gastrointestinal function. Classification of stool consistency using the Bristol Stool Chart. Numerical scale ranging from 1 (separate hard lumps) to 7 (liquid consistency with no solid pieces) with one-unit increments. Monitored longitudinally at months 0, 3, 15 and 27.
Gastrointestinal transit time | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome related to gastrointestinal function. Measurement of transit time through the digestive system using a so-called maize test. Participants consume 100 grams of sweet maize in the morning between 5.30-10.00 while still in a fasting state. The exact date and time of consumption is registered and so is the exact date and time when maize is observed for the first time in feces. Transit time is expressed as the difference between the ingestion and fecal excretion timepoints in hours. Monitored longitudinally at months 0, 3, 15 and 27.
Antibody-coating of fecal microbes | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome related to gastrointestinal function. Evaluation of endogenous antibody-coating of fecal microbes (bacteria, viruses etc) as well as the ability of fecal microbes to be bound by disease-related and other antibodies. Monitored longitudinally at months 0, 3, 15 and 27.
Fecal pH | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome related to gastrointestinal function. Monitored longitudinally at months 0, 3, 15 and 27.
Bacterial polysaccharides | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome related to gastrointestinal function. Lipopolysaccharide (LPS, endotoxin) and LPS-binding protein, capsular polysaccharides or other bacterial polysaccharides measured in blood samples as a biomarker of bacterial translocation across the intestinal epithelium. Monitored longitudinally at months 0, 3, 15 and 27.
Intestinal fatty acid binding protein | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome related to gastrointestinal function. Measurements of intestinal fatty acid binding protein in blood samples as a biomarker of enterocyte damage. Monitored longitudinally at months 0, 3, 15 and 27.
Pre-haptoglobin 2 | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome related to gastrointestinal function. Measurement of pre-haptoglobin 2 in blood samples as a biomarker of intestinal permeability. Monitored longitudinally at months 0, 3, 15 and 27.
Citrulline | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome related to gastrointestinal function. Measurement of citrulline in blood samples as a biomarker of intestinal function. Monitored longitudinally at months 0, 3, 15 and 27.
Calprotectin | The time between month 0 and month 27 after initiation of supplementation.
  Exploratory outcome related to gastrointestinal function. Calprotectin measured in fecal samples as a biomarker of intestinal inflammation. Monitored longitudinally at months 0, 3, 15 and 27.
Questionnaire-based self-reporting of experienced effects | The time between month 3 and month 27 after initiation of supplementation.
  A safety outcome. Study participants are asked whether they have experienced any positive or negative effects and whether they believe they have been given IPA or placebo. Evaluated at months 3, 12, 15, 24 and 27.
Registration of side effects | The time between month 0 and month 27 after initiation of supplementation.
  A safety outcome. Interviews with the aim of uncovering any side effects or adverse events. Results are registered using the REDCap instrument "CDISC|CDASHIG v2.1|Adverse Events". Evaluated at months 3, 12, 15, 24 and 27.
Leucocyte counts | The time between month 0 and month 27 after initiation of supplementation.
  A safety outcome. Total leucocytes, basophils, eosinophils, lymphocytes, monocytes, neutrophils as well as the joint group of metamyelo-, myelo- and promyelocytes. All counted in whole blood samples (x10^9/l). Monitored at months 0, 3, 15 and 27.
Thrombocytes | The time between month 0 and month 27 after initiation of supplementation.
  A safety outcome. Thrombocytes measured in whole blood (x 10^9/L). Monitored at months 0, 3, 15 and 27.
Hemoglobin | The time between month 0 and month 27 after initiation of supplementation.
  A safety outcome. Hemoglobin measured in whole blood (mmol/l). Monitored at months 0, 3, 15 and 27.
Alanine transaminase (ALT) | The time between month 0 and month 27 after initiation of supplementation.
  A safety outcome. Plasma alanine transaminase (ALT, U/l) measured as a biomarker of liver function. Monitored at months 0, 3, 15 and 27.
Aspartate aminotransferase (AST) | The time between month 0 and month 27 after initiation of supplementation.
  A safety outcome. Plasma aspartate aminotransferase (U/l) also known as aspartate transaminase measured as a biomarker of liver and muscle damage. Monitored at months 0, 3, 15 and 27.
Lactate dehydrogenase (LDH) | The time between month 0 and month 27 after initiation of supplementation.
  A safety outcome. Lactate dehydrogenase measured in plasma (U/l). Monitored at months 0, 3, 15 and 27.
Bilirubin | The time between month 0 and month 27 after initiation of supplementation.
  A safety outcome. Bilirubins measured in plasma (µmol/L) as a biomarker of liver function. Monitored at months 0, 3, 15 and 27.
Alkaline phosphatase | The time between month 0 and month 27 after initiation of supplementation.
  A safety outcome. Alkaline phosphatase (U/l) as a biomarker of liver function. Monitored at months 0, 3, 15 and 27.
Thyroid-stimulating hormone (TSH) | The time between month 0 and month 27 after initiation of supplementation.
  A safety outcome. Thyroid-stimulating hormone measured in plasma (mU/L) as a biomarker of thyroid function. Monitored at months 0, 3, 15 and 27.
Thyroxine (T4) | The time between month 0 and month 27 after initiation of supplementation.
  A safety outcome. Monitored in blood samples as a biomarker of thyroid function at months 0, 3, 15 and 27.
Triiodothyronine (T3) | The time between month 0 and month 27 after initiation of supplementation.
  A safety outcome. Monitored in blood samples as a biomarker of thyroid function at months 0, 3, 15 and 27.
Albumin | The time between month 0 and month 27 after initiation of supplementation.
  A safety outcome. Albumin measured in plasma (g/L). Monitored at months 0, 3, 15 and 27.
Coagulation factors II, VII and X (international normalized ratio (INR)) | The time between month 0 and month 27 after initiation of supplementation.
  A safety outcome. Coagulation factors II, VII and X (INR) measured in citrate plasma as a biomarker of coagulation. Monitored at months 0, 3, 15 and 27.
Creatinine | The time between month 0 and month 27 after initiation of supplementation.
  A safety outcome. Plasma creatinine (µmol/L) as a biomarker of kidney function. Monitored at months 0, 3, 15 and 27.
Estimated glomerular filtration rate (eGFR) | The time between month 0 and month 27 after initiation of supplementation.
  A safety outcome. Estimated glomerular filtration rate (eGFR/ 1,73m² (ml/min)) as a biomarker of kidney function. Monitored at months 0, 3, 15 and 27.
Counting of leftover capsules | The time between month 0 and month 27 after initiation of supplementation.
  A measure of compliance. Evaluated longitudinally at months 3, 12, 15, 24 and 27.
Questionnaire regarding demographic characteristics, socioeconomic background, lifestyle factors, and other potential confounding factors | The time between month 0 and month 24 after initiation of supplementation.
  Information on potential confounders or effect modifiers. The questionnaire is administered at months 0, 12 and 24.
Food frequency questionnaire | The time between month 0 and month 24 after initiation of supplementation.
  Information on potential confounders or effect modifiers. A food frequency questionnaire (FFQ) regarding dietary habits and food consumption during the past year is administered at months 0, 12 and 24.
Objective biomarkers of dietary intake | The time between month 0 and month 27 after initiation of supplementation.
  Information on potential confounders or effect modifiers. Measurement of fatty acids, vitamins, minerals, amino acids and food-derived DNA in blood, urine and fecal samples. Monitored at months 0, 3, 15 and 27.
Major Depression Inventory (MDI) | The time between month 0 and month 24 after initiation of supplementation.
  Information on potential confounders or effect modifiers. The Major Depression Inventory (MDI) score ranges from 0 to 50 with higher scores suggesting higher degrees of depression. Evaluated at months 0, 12 and 24.
Pittsburgh Sleep Quality Index (PSQI) | The time between month 0 and month 24 after initiation of supplementation.
  Information on potential confounders or effect modifiers. The global Pittsburgh Sleep Quality Index (PSQI) score is calculated. It ranges from 0 to 21 with higher scores indicating worse sleep quality. Evaluated at months 0, 12 and 24.

CONTACTS AND LOCATIONS:
Overall Officials: Jette Lautrup Frederiksen, MD, dr.med, professor, Principal Investigator — Copenhagen University Hospital, Rigshospitalet-Glostrup
Locations (1):
- Glostrup Hospital, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in published articles, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following publication of the article they are presented in.
Access Criteria: Researchers who provide a methodologically sound proposal can access the IPD to achieve the aims of the approved proposal. Proposals should be directed to jette.lautrup.battistini@regionh.dk. To gain access, data requestors will need to sign a data access agreement. Data and explanatory files will be made available at a third party website.